

# Statistical Analysis Plan

NCT Number: NCT04213209

Title: Specified drug use Surveillance for ADCETRIS Intravenous Infusion 50 mg
"Relapsed or refractory CD30 positive peripheral T-cell lymphoma and Hodgkin
lymphoma (pediatric only)"

Study Number: C25021

Document Version and Date: Version 2 / 21-Nov-2023

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

Takeda Pharmaceutical Company Limited Director, Biostatistics

Edition 2: Prepared on November 21, 2023

# TABLE OF CONTENTS

| 1 | Defin | nitio | ns of Terms, etc. | 3 |
|---|---|---|---|---|
| | | | of Terms and Abbreviations | 3 |
| | 1.2 | Ana | lysis Sets | 3 |
| | 1.3 | Nur | nber of digits to be displayed | 6 |
| | 1.4 | Imp | ortant identified risks, important potential risks, and important missing information | 7 |
| 2 | Num | ber | of study sites and patients enrolled and patient composition | ~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~ |
| | 9 1 | Dier | position of subjects | 8 |
| 3 | Patie | ent c | haracteristics | 9 |
| | 3.1 | Pati | ent characteristics | 9 |
| 4 | Deta | ils o | haracteristics | . 11 |
| | 4.1 | Adn | ninistration status of this drug | . 11 |
| 5 | Matt | ters 1 | related to safety | .12 |
| | 5.1 | Stat | tus of Occurrence of Adverse Events and Adverse Drug Reactions/Infections | |
| | 5.1 | 1.1 | Occurrence of adverse events | .12 |
| | 5.1 | 1.2 | Occurrence status of adverse reactions/infections | .12 |
| | 5.1 | 1.3 | Incidences of adverse events and adverse drug reactions/infections included in the safety | |
| | | | specifications | .13 |
| | 5.2 | | sus of occurrence of adverse events, adverse drug reactions, and infections in patients | |
| | | ex | cluded from safety evaluation | .14 |
| | 5.2 | 2.1 | Status of adverse events in patients excluded from safety evaluation | .14 |
| | 5.2 | 2.2 | Occurrence Status of Adverse Reactions/Infections in Patients Excluded from Safety | |
| | | | Evaluation | .15 |
| | 5.3 | Occ | urrence status of adverse events and adverse drug reactions/infections by seriousness, | |
| | | | ${\it CCAE~Grade~(worst~value), timing~of~onset, outcome, and~causal~relationship~with~this~drug}$ | .15 |
| | 5.3 | 3.1 | Occurrence of adverse events by seriousness, CTCAE Grade (worst value), timing of onset, | |
| | | < | outcome, and causal relationship with this drug | .15 |
| | 5.3 | 3.2 | Occurrence status of adverse drug reactions/infections by seriousness, CTCAE Grade | |
| • | rec | ) | (worst value), timing of onset, and outcome | .17 |
| ( | 5.4 | Ons | et status of adverse reactions/infections by patient background and treatment factors | .18 |
| | 5.4 | 4.1 | Onset status of adverse reactions/infections by patient background factor and treatment | |
| | | | details factor | |
| | | 4.2 | Occurrence Status of Adverse Reactions/Infections by Gender | |
| | 5.4 | | Occurrence Status of Adverse Reactions/Infections by Age Group | .20 |
| | 5.5 | | urrence Status of Adverse Events and Adverse Drug Reactions/Infections for which Action | |
| | | Ta | ken with this drug was Discontinuation | .20 |

| 5.5.1 Incidences of adverse events leading to discontinuation of this drug 20 | |
|---|---|
| 5.5.2 Occurrence Status of Adverse Reactions/Infections for which Action Taken with this drug | |
| was Discontinuation | .21 |
| 5.6 Status of administration of this drug by outcome at the onset of adverse reactions/infections | .22 |
| 5.7 Status of administration of this drug due to adverse reactions/infections included in the safety | 0) |
| specifications | .22 |
| 6 Efficacy | .24 |
| 6.1 Tumor response during the first 12 months of this drug therapy | |
| 6.2 Antitumor effect in 12 months from the start of this drug by patient demographics and | |
| treatment factors | .24 |
| 6.2.1 Antitumor effect in 12 months from the start of this drug by patient demographics and | |
| treatment factors (adult) | .24 |
| 6.2.2 Antitumor effect in 12 months from the start of this drug by patient demographics and | |
| treatment factors (children) | .26 |
| 6.3 Overall survival | .26 |
| 7 Occurrence Status of Adverse Reactions/Infections in Additional Pharmacovigilance Plan | .27 |
| 7.1 Incidences of ADRs and infections included in additional pharmacovigilance plan (Attached | |
| Form 12) | .27 |
| 8 Case Summary for Post-marketing Surveillance, etc. | .28 |
| 8.1 Case summary in post-marketing surveillance, etc. (Attached Form 16) | |
| Preparation history (version control) | .29 |
| [Appendix 1] Comparison table of changes | 1 |
| Property of Takeda. For non-cornine | |

### 1 Definitions of Terms, etc.

### 1.1 List of Terms and Abbreviations

- This drug: Adcetris for Intravenous Drip Infusion 50 mg is abbreviated as this drug.
- Adverse Event: AE occurred after administration of this drug.
- Adverse reactions, etc.: An abbreviation for the term "adverse reactions/infections." Adverse events that are not "not related" to this drug as assessed by the managing physician. This statistical analysis plan uses "adverse drug reactions/infections" in the title and "adverse drug reactions, etc." in the text and tables.
- Serious adverse events: Adverse events assessed as "serious" by the investigator. Using the Important Medical Events
   List, events listed in the MedDRA code list (PT code) will be handled as serious even if the investigator's assessment is "non-serious."
- Related to this drug: An AE that is not related to this drug.
- Not related to this drug: An AE that is not related to this drug.
- Summary statistics: A collective term for sample size, mean, standard deviation, maximum, minimum, and quartiles.
- Patients whose CRFs were not collected: Registered patients whose CRFs were not collected.
- Patients whose CRFs were collected: Registered patients whose CRFs were collected.
- Days after administration: Day -1 is defined as the day before the start date of this drug treatment and Day 1 is defined as the start date of this drug treatment.
- Duration of treatment with this drug (days): The end date of treatment with this drug the start date of treatment with this drug +1
- Children: Patients aged < 18 years at the start of treatment.
- Adults: Patients aged 18 years or older at the start of treatment.
- Timing of onset of an adverse event (or adverse drug reaction, etc.): Calculated as the date of onset of the adverse event (or adverse drug reaction, etc.) the start date of the first dose of this drug +1.
- Duration of disease:
  - Actual number (months) = (Year of the first administration of this drug Year of the diagnosis of peripheral T-cell lymphoma or Hodgkin's lymphoma) ×12+ (Month of the first administration of this drug Month of the diagnosis of peripheral T-cell lymphoma or Hodgkin's lymphoma)
    - If the month of diagnosis is unknown, it should be calculated as January of the year of diagnosis.
- Time from the last day of treatment immediately before administration of this drug to the first administration of this drug (days): The first day of administration of this drug the last day of treatment immediately before administration of this drug +1

- BMI (kg/m<sup>2</sup>): Calculated as weight (kg)/height (m)<sup>2</sup> (rounded to the first decimal place).

- properly of Takeda. For non-commercial use only and subject to the applicable of takeda.

#### 1.2 **Analysis Sets**

Patients receiving this drug who had no major protocol violations and whose safety could be evaluated."

Specifically, patients with locked CRFs who meet any of the following criteria will be excluded from the safety analysis set.

This drug naïve

Presence/absence of adverse event unknown

Withdrawal of consent As the analysis population of the general drug use-results survey, the "subjects for safety evaluation" and the "subjects for

Siblicaple resi

Patients eligible for efficacy evaluation

In this statistical analysis plan, the "Patients evaluable for efficacy with no major protocol deviations among patients evaluated for safety" will be defined as the patients evaluated for efficacy. Patients who meet the following conditions among the patients evaluated for safety will be excluded from the patients evaluated for efficacy.

- · Other than target disease [revealed after the fact]
- Violation of inclusion criteria [revealed after the fact]
- r than target disease [revealed after the fact]
  ation of inclusion criteria [revealed after the fact]

  Patients who do not meet the following inclusion criteria will be excluded from the efficacy analysis set as violation of the inclusion criteria.
  - Patients with relapsed or refractory disease
- ve for CD3

  ve for CD3

  roperty of Takeda.

  For non-commercial

  Property of Takeda. Patients who are positive for CD30

Property of Takeda. For non-commercial use only and subject to the applicable Temes of use

- Properly of Takeda. For non-commercial use only and subject to the applicable Tames of use

# Number of study sites and patients enrolled and patient composition

#### 2.1 Disposition of subjects

Analysis population: Specified use-results survey

Analysis population: All enrolled patients (patients enrolled)

Analysis item: Patients enrolled

Medical institution inspected

CRF not collected

CRF collected

counting)

Patients excluded from safety evaluation

Reason for exclusion (multiple

oplicable terms of Use [this drug was not administered, presence or absence of

adverse events was unknown, and consent was

withdrawn.]

Subjects evaluable for safety

Patients excluded from efficacy

evaluation '

Reason for exclusion (multiple

[Other than the target disease [Found after the fact],

counting)

Violation of inclusion criteria [found out after the

fact]

Patients eligible for efficacy evaluation

#### 3 **Patient characteristics**

#### 3.1 **Patient characteristics**

Analysis population: Subjects evaluable for safety

Gender [Male, female] Analysis item:

[Min <= - < 18, 18 <= - < 30, 30 <= - < 40, 40 Age (years)

Disease duration (months)

[Peripheral T-cell lymphoma (PTCL), Hodgkin Diagnosis

[Peripheral T-cell lymphoma not otherwise Type of PTCL

specified (PTCL-NOS), angioimmunoblastic

T-cell lymphoma (AITL), adult T-cell

leukemia/lymphoma (ATLL), ALK-positive

anaplastic large cell lymphoma (ALK+

ALCL) [for patients aged < 18 years], ALK-

negative anaplastic large cell lymphoma

(ALK-ALCL) [for patients aged < 18 years],

other]

(details on adult T-cell leukemia/lymphoma

[Acute type, lymphoma type, others]

[ATLL])

Disease site (multiple counting) [Lymph nodes, spleen, liver, lung, bone, CNS,

bone marrow, skin, others]

[Stage I, II, III, IV, unknown]

[Stage I, II, III, IV, unknown]

Clinical stage

Ann Arbor Classification

Murphy classification

Presence or absence

Relapsed/ref

ECC Presence or absence of B symptoms [Absent, present]

[Relapsed/refractory]

[0, 1, 2, 3, 4]

Treatment category (at the start of this drug

[Outpatient/inpatient]

[Absent, present]

Presence or absence of medical history [Absent, present, unknown]

[Never smoked, current smoker, former smoker

Smoking history but not current smoker, unknown] Weight (kg) [Min <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - <

60.0, 60.0<= - < 70.0, 70.0 <= - <= Max, not

BMI(kg/m2)

Pregnancy (females only)

Breastfeeding status (females only)

Treatment for PTCL or HL before the start of this

drug

Number of regimens

[0, 1, 2, 3, 4, ≥ 5, unknown]

[(1) A+CHP, (2) CHOP, (2)

(5) GDP, (4)

oth Drug therapy

others, unknown]
[Absent, present, unknown] Radiotherapy

[Absent, present, unknown] Hematopoietic stem cell transplantation

[Autologous transplant, allogeneic transplant]

...t) [Au
...ent immediately
...n of this drug to the first
...on of this drug (days)
...above analytical variables, frequency tabulation of d
continuous data will be calculated. This tabulation will be per
(PTCL-NOS, ATPL, ATLL, others) and children (PTCL, HL). For the above analytical variables, frequency tabulation of discrete data and summary statistics of continuous data will be calculated. This tabulation will be performed for cases of overall, adults

# **Details of treatment**

#### 4.1 Administration status of this drug

Analysis population: Subjects evaluable for safety

Analysis item: This drug loading dose (mg/kg)

 $\begin{array}{l}
 < 1.2, 1.2 <= - < 1.8, 1.8, \\
 < 1.0 < - <= Max] \\
[Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <= - < 1.8, 1.8, \\
 < 1.8 < - <= Max] \\
[Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <- \\
 < 1.8 < - <= M
\end{array}$ Mean dose of this drug per administration

(mg/kg)

This drug dose per 3 weeks (mg/kg/3 weeks)

[1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17] Maximum number of doses

Reasons for Discontinuation of this drug

(Multiple Count)

[The treatment goal was achieved, the patient did

not visit the hospital due to the onset of adverse

events, transfer to another hospital, etc.,

pregnancy, disease progression, hematopoietic

stem cell transplantation, follow-up

observation, patient's or family's wish, etc.]

For the above analytical variables, frequency tabulation of discrete data and summary statistics of Analytical method:

continuous data will be calculated. This tabulation will be performed for cases of overall, adults

Property of Takeda. For non-commercial (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL).

# Matters related to safety

#### 5.1 Status of Occurrence of Adverse Events and Adverse Drug Reactions/Infections

#### 5.1.1 Occurrence of adverse events

Analysis population:

Analysis item:

une above analytical variable, the following analyses should be performed. This tabulation will be performed for all patients, adults (PTCL-NOS, AITL, ATLL, others), and children (PTCL, HL).

(1) Number of subjects with adverse events

(2) Number of AEs

(3) Incidence of adverse events

(4) T-Analytical method: applicable applicable

- (4) Type of Adverse Event

The calculation method for each analysis is as follows.

[Number of subjects with adverse events]

Number of patients with adverse events.

[Number of adverse events]

Number of AEs that occurred. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

Calculated as the number of patients with adverse events/number of patients evaluated for safety ×100.

[Type of adverse event]

- AEs will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
  - Within SOC, the number of patients with adverse events and the incidence rate will be described using internationally agreed SOC order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.
- By PT, the number of patients with adverse events and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.

# Occurrence status of adverse reactions/infections

Subjects evaluable for safety

Adverse reactions, etc.

For the above analytical variable, the following analyses should be performed. This tabulation will

be performed for cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL,

HL).

- (1) Number of patients with adverse reactions, etc.
- (2) Number of adverse drug reactions
- (3) Incidence of adverse drug reactions
- (4) Types of adverse reactions, etc.

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions]

• Number of patients with adverse reactions, etc.

[Number of adverse reactions]

Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc.
 occurs multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions]

- Number of patients with adverse drug reactions/Number of patients evaluated for safety ×100.
   [Types of adverse reactions, etc.]
- Adverse drug reactions will be coded using MedDRA/JOI will be roughly classified by SOC
  and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in
  ascending order of HLGT code, but do not output) and PT.
- In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be
  described in SOC internationally agreed order. A subject with multiple occurrences of an
  event within an SOC should be counted only once for that SOC.
- By PT, the number of patients with adverse drug reactions, etc. and the incidence will be
  described in ascending order of PT codes. A subject who experienced the same PT more than
  once should be counted as 1 subject with the PT.

# 5.1.3 Incidences of adverse events and adverse drug reactions/infections included in the safety specifications

# 5.1.3.1 Incidences of adverse events included in the safety specifications

Analysis population: Subjects evaluable for safety

Analysis item: Adverse events included in the safety specifications (important identified risks)

Stratification item: Seriousness [Serious, non-serious]

Analytical method: For the above analysis set, analyses should be performed in the same manners as in Section 5.1.1

for each risk and each stratum of the stratification factor. This tabulation will be performed for

cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL). A subject who

experienced the same SOC/PT more than once should be counted as 1 subject in the SOC/PT.

However, if the seriousness differs, 1 subject will be counted for each of serious and non-serious.

The target risks shall follow the definitions described in the important identified risks.

# 5.1.3.2 Incident Status of Adverse Reactions/Infections Included in Safety Specifications

Analysis population: Subjects evaluable for safety

Analysis item: Adverse reactions, etc. corresponding to safety specifications (important identified risks)

Stratification item: Seriousness [Serious, non-serious]

Analytical method:

# Status of occurrence of adverse events, adverse drug reactions, and infections in patients excluded from safety 5.2 evaluation

#### 5.2.1 Status of adverse events in patients excluded from safety evaluation

Analysis population: Patients excluded from safety evaluation

Analysis item: Adverse Events

For the above analytical variable, the following analyses should be performed. Analytical method:

(1) Number of subjects with adverse events

- (2) Number of AEs
- Incidence of adverse events
- (4) Type of Adverse Event

The calculation method for each analysis is as follows.

[Number of subjects with adverse events]

Number of patients with adverse events.

Number of AEs that occurred. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

Number of patients with adverse events/Number of patients excluded from safety evaluation

- Number of AEs that c
  patient, the total numb
  [Incidence of adverse events]

  Number of patients with
  ×100.

  [Type of adver• AEs will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
  - Within SOC, the number of patients with adverse events and the incidence rate will be described using internationally agreed SOC order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.

By PT, the number of patients with adverse events and the incidence will be described in 3ct to the applicable Terms of Use ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.

#### 5.2.2 Occurrence Status of Adverse Reactions/Infections in Patients Excluded from Safety Evaluation

Analysis population: Patients excluded from safety evaluation

Analysis item: Adverse reactions, etc.

Analytical method: For the above analytical variable, the following analyses should be performed.

- (1) Number of patients with adverse reactions, etc.
- (2) Number of adverse drug reactions
- Incidence of adverse drug reactions
- Types of adverse reactions, etc.

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions, etc.]

Number of patients with adverse reactions, etc.

[Number of adverse reactions]

Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions, etc.]

Number of patients with adverse drug reactions/Number of patients excluded from safety evaluation ×100.

[Types of adverse reactions, etc.]

Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.

In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.

- By PT, the number of patients with adverse drug reactions, etc. and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.
- Occurrence status of adverse events and adverse drug reactions/infections by seriousness, CTCAE Grade (worst value), timing of onset, outcome, and causal relationship with this drug
- Occurrence of adverse events by seriousness, CTCAE Grade (worst value), timing of onset, outcome, and causal relationship with this drug

Subjects evaluable for safety Analysis population:

Analysis item: Adverse Events

Stratification item: Total

Seriousness [Serious, non-serious]

CTCAE Grade (worst value) [Grade1, Grade2, Grade3, Grade4, Grade5]

Timing of onset (day)  $[1 \le - \le 21, 22 \le - \le 84, 85 \le - \le 168, 169]$ 

<= - <= 252, 253 <= - <= 336, 337 <= - <= Max]

Timing of onset (number of doses) [From after the 1st dose to before the 2nd dose, from

after the 2nd dose to before the 5th dose, from after the 5th dose to before the 9th dose, from after the 9th dose to before the 13th dose, from after the 13th dose to before the 17th dose, from

after the 17th dose]

Outcome [Recovered/resolved, resolving, not recovered,

recovered with sequelae, fatal (due to this event),

unknown]

Relationship to this drug [Related, Not Related]

Analytical method: For the above analysis set, analyses similar to those in Section 5.1.1 will be performed for each

stratum of the stratification factor. This tabulation will be performed for cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL). A subject who experienced the same SOC/PT more than once should be counted as 1 subject in the SOC/PT. However, 1 subject within the same SOC will be included in the study according to the following order of priority, and 1

subject within the same PT will be included in the study according to the following order of priority for any of the stratification factors.

Seriousness: Serious → Non-serious

CTCAE Grade (worst value): Grade5→Grade4→Grade3→Grade2→Grade1

Timing of onset (days): 1 to 21 days  $\rightarrow$ 22 to 84 days  $\rightarrow$ 85 to 168 days  $\rightarrow$ 169 to 252 days  $\rightarrow$ 253 to

336 days  $\rightarrow \ge 337$  days

Timing of onset (number of doses): After the first dose to before the second dose  $\rightarrow$  After the second dose to before the fifth dose  $\rightarrow$  After the fifth dose to before the ninth dose  $\rightarrow$  After the ninth dose to before the thirteenth dose  $\rightarrow$  After the thirteenth dose to before the seventeenth dose

→ After the seventeenth dose and thereafter

Outcome: Death (due to this event)  $\rightarrow$  recovered with sequelae  $\rightarrow$  not recovered  $\rightarrow$  recovering  $\rightarrow$ 

recovered → unknown

Property of Lakedai. For

Causal relationship with this drug: Related → Not related

#### 5.3.2 Occurrence status of adverse drug reactions/infections by seriousness, CTCAE Grade (worst value),

# timing of onset, and outcome

Analysis population: Subjects evaluable for safety

Adverse reactions, etc. Analysis item:

Stratification item: Total

> Seriousness [Serious, non-serious]

[Grade1, Grade2, Grade3, Grade4, Grade5] CTCAE Grade (worst value)

Terms of Use [1 <= - <= 21, 22 <= - <= 84, 85 <= - <= 168, 169 Timing of onset (day)

<= - <= 252, 253 <= - <= 336, 337 <= 7 <= Max]

[From after the 1st dose to before the 2nd dose, from Timing of onset (number of doses)

> after the 2nd dose to before the 5th dose, from after the 5th dose to before the 9th dose, from after the 9th dose to before the 13th dose, from after the 13th dose to before the 17th dose, from

after the 17th dose onwards]

[Recovered/resolved, resolving, not recovered, Outcome

recovered with sequelae, fatal (due to this event),

unknown]

Analytical method:

Property of Lakeda. For

For the above analysis set, analyses similar to those in Section 5.1.2 will be performed for each stratum of the stratification factor. This tabulation will be performed for cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL). A subject who experienced the same SOC/PT more than once should be counted as 1 subject in the SOC/PT. However, 1 subject within the same SOC will be included in the study according to the following order of priority, and 1 subject within the same PT will be included in the study according to the following order of priority for any of the stratification factors.

Seriousness: Serious → Non-serious

CTCAE Grade (worst value): Grade5→Grade4→Grade3→Grade2→Grade1

Timing of onset (days): 1 to 21 days  $\rightarrow$ 22 to 84 days  $\rightarrow$ 85 to 168 days  $\rightarrow$ 169 to 252 days  $\rightarrow$ 253 to 336 days →  $\ge$  337 days

Timing of onset (number of doses): After the first dose to before the second dose → After the second dose to before the fifth dose  $\rightarrow$  After the fifth dose to before the ninth dose  $\rightarrow$  After the ninth dose to before the thirteenth dose - After the thirteenth dose to before the seventeenth dose → After the seventeenth dose and thereafter

Outcome: Death (due to this event) → recovered with sequelae → not recovered → recovering → recovered → unknown

# Onset status of adverse reactions/infections by patient background and treatment factors

#### 5.4.1 Onset status of adverse reactions/infections by patient background factor and treatment details factor

Analysis population: Subjects evaluable for safety

Analysis item: Adverse reactions, etc.

Stratification item: [Male, female] Gender

> [Min <= - < 18, 18 <= - < 30, 30 <= - < 40, 40 Age (years)

[Peripheral T-cell lymphoma (PTCL), Hodgkin Diagnosis

lymphoma (HL)]

[Peripheral T-cell lymphoma not otherwise Type of PTCL

specified (PTCL-NOS), angioimmunoblastic

T-cell lymphoma (AITL), adult T-cell

leukemia/lymphoma (ATLL), ALK-positive

Sanaplastic large cell lymphoma (ALK+

ALCL) [for patients aged < 18 years], ALK-

negative anaplastic large cell lymphoma

(ALK-ALCL) [for patients aged < 18 years],

other]

[Acute type, lymphoma type, others]

[Lymph nodes, spleen, liver, lung, bone, CNS,

bone marrow, skin, others]

n
(A
othe

(details on adult T-cell leukemia/lymphoma

ATLL])
sease site (multiple counting)

'al stage

Arber Ann Arbor Classification [Stage I, II, III, IV, unknown]

Murphy classification [Stage I, II, III, IV, unknown]

Clinical stage
Ann Arbor C'
Murph
P Presence or absence of B symptoms [Absent, present] Relapsed/refractory status [Relapsed/refractory]

**ECOG Performance Status** [0, 1, 2, 3, 4]

Treatment category (at the start of this drug

[Outpatient/inpatient]

[Absent, present]

Presence or absence of medical history [Absent, present, unknown] Weight (kg) [Min <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - <

60.0, 60.0<= - < 70.0, 70.0 <= - <= Max, not

measured]

BMI(kg/m2) [Min <= - < 18.5, 18.5 <= - < 25.0, 25.0 <= - <

 $30.0, 30.0 \le - \le Max$ 

Treatment for PTCL or HL before the start of this

drug

[(1) A+CHP, (2) CHOP, (3) ABVD, (4) mLSG15, Drug therapy

(5) GDP, (6) OEPA/OPPA,

others, unknown]

[Absent, present, unknown] Radiotherapy

Hematopoietic stem cell transplantation [Absent, present, unknown]

(With haematopoietic stem cell transplant) [Autologous transplant, allogeneic transplant]

Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <= - < 1.8, 1.8, 1.8 < - <= Max1 This drug loading dose (mg/kg)

Mean dose of this drug per administration [Min  $\leq$  - < 0.9, 0.9  $\leq$  - < 1.2, 1.2  $\leq$  - < 1.8,

1.8, 1.8 < - <= Max(mg/kg)

This drug dose per 3 weeks (mg/kg/3 weeks) [Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <= - < 1.8,

1.8, 1.8 < - <= Max

For the above analytical variable, the following analyses will be performed for each stratum of the Analytical method:

stratification factor. This tabulation will be performed for cases of overall, adults (PTCL-NOS,

AITL, ATLL, others) and children (PTCL, HL).

Number of patients with adverse reactions, etc.

Incidence of adverse drug reactions

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions]

Number of patients with adverse reactions, etc.

[Incidence of adverse reactions]

Number of patients with adverse drug reactions/Number of patients evaluated for safety ×100.

# Occurrence Status of Adverse Reactions/Infections by Gender

Analysis population: Subjects evaluable for safety

Adverse reactions, etc.

[Male, female] Gender

For the above analysis set, analyses similar to those in Section 5.1.2 will be performed for each Analytical method:

stratum of the stratification factor. This tabulation will be performed for cases of overall, adults

(PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL).

#### 5.4.3 Occurrence Status of Adverse Reactions/Infections by Age Group

Analysis population: Subjects evaluable for safety

Analysis item: Adverse reactions, etc.

[Min <= - < 12, 12 <= - < 18, 18 <= - < 30, Stratification item: Age (years) (all subjects)

[Min <= - < 18, 18 <= - < 30, 30 <= - < 40, Age (years) (adult)

Age (years) (children)

For the above analysis set, analyses similar to those in Section 5.1.2 will be performed for each Analytical method:

stratum of the stratification factor. This tabulation will be performed for cases of overall, adults

(PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL).

# Occurrence Status of Adverse Events and Adverse Drug Reactions/Infections for which Action Taken with this 5.5 drug was Discontinuation

#### Incidences of adverse events leading to discontinuation of this drug 5.5.1

Analysis population: Subjects evaluable for safety

AEs leading to discontinuation of this drug Analysis item:

For the above analytical variable, the following analyses should be performed. This tabulation will Analytical method: Property of Lakeda. For

be performed for all patients, adults (PTCL-NOS, AITL, ATLL, others), and children (PTCL, HL).

- Number of patients with adverse events leading to discontinuation of this drug
- Number of AEs leading to this drug discontinuation
- Incidence of AEs leading to discontinuation of this drug
- Adverse event type for which action taken with this drug was discontinuation

The calculation method for each analysis is as follows.

[Number of patients with adverse events for which this drug treatment was discontinued]

Number of subjects with AEs leading to discontinuation of this drug.

[Number of adverse events for which this drug was discontinued]

Number of adverse events for which the action taken with this drug was discontinuation. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events for which action taken with this drug was discontinuation]

Calculate the number of patients with adverse events whose action taken with this drug is discontinuation/the number of patients included in the safety evaluation  $\times 100$ .

[Action taken with this drug was treatment discontinuation due to type of adverse event]

- erms of Use AEs leading to discontinuation of this drug will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- For SOC, the number of patients with adverse events whose action taken with this drug is treatment discontinuation and the incidence are described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.
- By PT, the number of patients with adverse events whose action taken with this drug was treatment discontinuation and the incidence thereof will be entered in ascending order of PT code. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.

#### 5.5.2 Occurrence Status of Adverse Reactions/Infections for which Action Taken with this drug was

# Discontinuation

Subjects evaluable for safety Analysis population:

Adverse reactions, etc. for which the action taken with this drug is discontinuation of administration Analysis item: For the above analytical variable, the following analyses should be performed. This tabulation will Analytical method: be performed for cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL,

HL).

- (1) Number of patients with adverse drug reactions, etc. for which this drug treatment was discontinued
- Number of ADRs leading to discontinuation of this drug
- Incidence of adverse drug reactions/infections leading to discontinuation of this drug
- Type of adverse drug reaction, etc. for which action taken with this drug is discontinuation The calculation method for each analysis is as follows.

[Number of patients with adverse drug reactions, etc. for which this drug was discontinued]

- Action taken with this drug was number of patients with adverse drug reactions. [Action taken with this drug was number of adverse drug reactions requiring treatment discontinuation]
- Property of Takeda. For no (2)
  (3) Number of adverse drug reactions, etc. for which action taken with this drug was discontinuation. If the same adverse drug reaction, etc. occurs multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse drug reactions, etc. for which treatment with this drug was discontinued]

Calculate the number of patients with adverse drug reactions, etc. for which actions taken for this drug are discontinuation/the number of patients included in the safety evaluation  $\times 100$ .

[Action taken with this drug was treatment discontinuation due to type of adverse reactions, etc.]

- Adverse drug reactions, etc. for which this drug treatment is discontinued will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- In SOC, the number of patients with adverse drug reactions, etc. for which the action taken with this drug is treatment discontinuation and the incidence are described in SOC? internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.
- By PT, action taken with this drug was treatment discontinuation Describe the number of patients with adverse reactions, etc. and the incidence in ascending order of PT code. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.

#### Status of administration of this drug by outcome at the onset of adverse reactions/infections 5.6

Analysis population: Subjects evaluable for safety

Analysis item: Number of adverse drug reactions

Stratification item 1: Presence or absence of changes due to this event [Absent, present]

[Dose reduction, dose interruption [dose delay],

Details of changes (duplicate counting) [\*] [\*]

discontinuation]

Stratification item 2: [Recovered/resolved, resolving, not recovered,

recovered with sequelae, fatal, unknown]

Analytical method: For the above analysis set, the number of adverse drug reactions, etc. will be tabulated for each stratum of Stratification Item 1 and the number of events will be tabulated for each stratum of Stratification Item 2. This tabulation will be performed for cases of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL). The denominator for the incidence rate per Stratum Item 1 will be the number of events per stratum in Stratum Item 2.

# Status of administration of this drug due to adverse events and adverse drug reactions/infections included in the safety specifications

# Administration status of this drug due to adverse events included in the safety specifications

Analysis population: Subjects evaluable for safety

Adverse events included in the safety specifications (Important identified risks: peripheral neuropathy, Analysis item:

bone marrow depression)

Stratification item: Presence or absence of changes due to this event [Absent, present]

> Details of changes (duplicate counting) [Dose reduction, dose interruption [dose delay],

> > discontinuation]

Analytical method: For the above analysis subjects, the number of adverse events will be tabulated by frequency by

insofuse CTCAE Grade (worst value) of adverse events falling under each risk and stratified by stratification item. For the incidence rate for each stratification factor, the denominator will be the number of events for each CTCAE Grade (worst value). This tabulation will be performed for cases of overall, adults

(PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL).

#### 5.7.2 Status of administration of this drug due to adverse reactions/infections included in the safety

# specifications

Analysis population: Subjects evaluable for safety

Adverse reactions, etc. corresponding to safety specifications (Important identified risks: peripheral Analysis item:

neuropathy, bone marrow depression)

Presence or absence of changes due to this event Stratification item: [Absent, present]

> Details of changes (duplicate counting) [Dose reduction, dose interruption [dose delay],

> > discontinuation]

Analytical method: In the above analysis population, the number of adverse drug reactions, etc. will be tabulated for

frequency by stratification item by CTCAE Grade (worst value) of adverse drug reactions, etc.

corresponding to each risk. For the incidence rate for each stratification factor, the denominator will be the number of events for each CTCAE Grade (worst value). This tabulation will be performed for cases

an of overall of takeda. For non-co of overall, adults (PTCL-NOS, AITL, ATLL, others) and children (PTCL, HL).

# **Efficacy**

#### 6.1 Tumor response during the first 12 months of this drug therapy

Analysis population: Patients whose antitumor effect was assessed among the patients evaluated for efficacy

Analysis item: Antitumor effect

applicable Terms of Use [With PET assessment, without PET assessment, Stratification item: PTCL or HL other than adult T-cell

leukemia/lymphoma (ATLL) total]

\*Data will be tabulated in adults (PTCL-NOS, AITL, others), and children (PTCL, HL) and

separately.

ATLL

[For PTCL, For HL] Pediatric PTCL or HL (JPLSG version)

For each of the above analysis items, the frequency of assessment results will be tabulated for each Analytical method:

stratum of the stratification item in patients whose antitumor effect has been assessed among the

patients evaluated for efficacy, and the response rate will be calculated. In addition, a band graph will

be prepared for the above analysis results.

#### Antitumor effect in 12 months from the start of this drug by patient demographics and treatment factors 6.2

# 6.2.1 Antitumor effect in 12 months from the start of this drug by patient demographics and treatment factors (adult)

Patients whose antitumor effect was assessed among the patients evaluated for efficacy (adults) Analysis population:

Analysis item: Antitumor effect

PTCL or HL other than adult T-cell Stratification item 1: [With PET assessment, without PET assessment,

> leukemia/lymphoma (ATLL) total]

\*To be tabulated separately for PTCL-NOS,

AITL, and others

ATLL

Stratification item 2 Property of Lakeda. Gender [Male, female]

|Min| < - < 18, 18 < - < 30, 30 < - < 40, 40Age (years)

<= - < 50, 50 <= - < 60, 60 <= - < 70, 70 <= -

< 80, 80 <= - <= Max

[Peripheral T-cell lymphoma (PTCL), Hodgkin Diagnosis

lymphoma (HL)]

Type of PTCL [Peripheral T-cell lymphoma not otherwise

specified (PTCL-NOS), angioimmunoblastic

T-cell lymphoma (AITL), adult T-cell

leukemia/lymphoma (ATLL), ALK-positive

anaplastic large cell lymphoma (ALK+ ALCL) [for patients aged < 18 years], ALK-Terms of Use negative anaplastic large cell lymphoma (ALK-ALCL) [for patients aged < 18 years], other]

(details on adult T-cell leukemia/lymphoma

[Acute type, lymphoma type, others]

[ATLL])

[Lymph nodes, spleen, liver, lung, bone, CNS, Disease site (multiple counting)

bone marrow, skin, others]

Clinical stage

[Stage I, II, III, IV, unknown] Ann Arbor Classification [Stage I, II, III, [V] unknown] Murphy classification

Presence or absence of B symptoms [Absent, present]

[Relapsed/refractory] Relapsed/refractory status

**ECOG Performance Status** [0, 1, 2, 3, 4]

Treatment category (at the start of this drug [Outpatient/inpatient]

treatment)

[Absent, present] Complications Presence or absence of medical history

Weight (kg) |Min| <= - < 40.0, 40.0 <= - < 50.0, 50.0 <= - <

Treatment for PTCL or HL before the start of this drug

Number of regimens

Drug therapy 60.0, 60.0<= - < 70.0, 70.0 <= - <= Max, not

measured]

[Min <= - < 18.5, 18.5 <= - < 25.0, 25.0 <= - <

 $30.0, 30.0 \le - \le Max$ 

[Absent, present, unknown]

 $[0, 1, 2, 3, 4, \ge 5, unknown]$ 

[(1) A+CHP, (2) CHOP, (3) ABVD, (4) mLSG15,

(5) GDP, (6) OEPA/OPPA, (7) ALCL99,

others, unknown]

[Absent, present, unknown]

[Absent, present, unknown]

(With haematopoietic stem cell transplant) [Autologous transplant, allogeneic transplant] This drug loading dose (mg/kg)  $[Min \le - < 0.9, 0.9 \le - < 1.2, 1.2 \le - < 1.8,$ 

1.8, 1.8 < - <= Max

[Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <= - < 1.8, Mean dose of this drug per administration

1.8, 1.8 < - <= Max(mg/kg)

[Min <= - < 0.9, 0.9 <= - < 1.2, 1.2 <= - < 1.8, This drug dose per 3 weeks (mg/kg/3 weeks)

1.8, 1.8 < - <= Max

For each of the above analysis items, frequency will be tabulated by stratification item 1 and then by Analytical method:

stratum of stratification item 2 in patients (adults) whose antitumor effect has been assessed among

the efficacy evaluation set.

Antitumor effect in 12 months from the start of this drug by patient demographics and treatment factors 6.2.2

(children)

Efficacy analysis set with tumor response assessment (children) Analysis population:

Antitumor effect Analysis item:

[With PET assessment, without PET assessment, Stratification item 1: PTCL

HL

[With PET assessment, without PET assessment,

Pediatric PTCL or HL (JPLSG version) [For PTCL, For HL]

Analytical method: For each of the above analysis items, data will be tabulated in the same manner as in Section 6.2.1

in patients (children) whose antitumor effect has been assessed among the efficacy evaluation set,

stratified by stratification item 1.

6.3 Overall survival

Patients eligible for efficacy evaluation Analysis population:

Overall survival Analysis item:

Property of Lakeda. Analytical method: < For the above analysis set, the survival rate at 12 months will be estimated by the Kaplan-Meier

method, and Kaplan-Meier plots will be prepared. This tabulation will be performed for cases of

overall, adults (PTCL-NOS, AITL, ATLL, others), and children (PTCL, HL).

...ce Plan
...dee plan (Attached Form 12)
...predifications (important identified risks)
[Serious, row-serious]
...de following analyses should be performed for each of the autono in somethic with Oxtop 1-4 in Attached Form 12 to
...de No. 0322-10 dated Market 25, 2020.
...patients with events and insidence
...escription of risk names and risk names shall follow the definitions of the control of the autonomic risks and insidence
...escription of risk names and risk names shall follow the definitions of the control of the cont

# Case Summary for Post-marketing Surveillance, etc.

# some's some's applicable terms of Use 8.1 Case summary in post-marketing surveillance, etc. (Attached Form 16)

Analysis population: CRF collected

Analysis item: Case No.

Name of medical institution

Gender

Age

Reason for use (Disease code, disease name)

Comorbidity (Disease code, disease name)

Maximum dose

Route of administration

Mean dose

Unit

Duration of use (duration of this drug treatment)

Concomitant medications (Drug code, drug name)

Degree of effect

Adverse reactions (Disease code, disease name, outcome) CRF No.

Dropout

Reason for dropout

Name of disease (other than target disease)

A list of the above analysis items will be prepared in accordance with the reexamination data entry Analytical method:

file preparation guideline specified in the Notification No. 1119 (3) of the Pharmaceutical

Property of Takeda. For non-co Evaluation Division, PSEHB dated November 19, 2020.

| Version | Date | Author/Reporter | Comments |
|---|---|---|---|
| Original<br>Version | 2023.10.30 | | Preparation of initial version |
| Version 2 | 2023.11.21 | | Version 2 prepared |
| | | | Changes from Version 1 are described in Appendix 1. |

Property of Takeds. For non-commercial use only and subject to the applicable Temps of use

# [Appendix 1] Comparison table of changes

Statistical Analysis Plan (Version 1, prepared on October 30, 2023 → Version 2, prepared on 21/11/2023)

| Statistical Linery | any sist 1 min ( version 1; prepared on George 30; 2023 · version 2; prepared on 21/11/2023) | | |
|---|---|---|---|
| Page | Before amendment | After amendment | Reason for change |
| 22 | | 5.6 Status of this drug administration by outcome at the | Description adjustment. |
| | | onset of adverse drug reactions/infections | |
| | | Addition of description about the incidence rate | |
| 22 | | 5.7 Status of administration of this drug due to adverse | Due to addition of tabulation. |
| | | events and adverse drug reactions/infections included in | |
| | | the safety specifications | |
| | | Item added | |



